CLINICAL TRIAL: NCT06243601
Title: Effect of Aloe Vera Gel as an Intra Canal Medicament in Patients With Asymptomatic Periapical Lesions.
Brief Title: Effect of Aloe Vera Gel as an Intra Canal Medicament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IslamabadDentalHospital
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Periapical Diseases
Keywords: Antibacterial, Analgesic, Clinical signs and symptoms
MeSH Terms: conditions — Periapical Diseases; Signs and Symptoms | interventions — Aloe vera gel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Fresh AVG will be prepared. It will be placed as intracanal medicament after cleaning and shaping in patients with asymptomatic periapical lesions
  Interventions: Biological: Aloe vera Gel
- Control Group (No Intervention): No intracanal medicament will be placed

INTERVENTIONS:
Biological: Aloe vera Gel — A fresh aloe vera (Aloe Barbadensis) leaf will be plucked from the plant. The leaf will be washed with normal saline, peeled with scalpel and the inner gel will be blended in a blender to convert it into a watery consistency. The solution will be stored in an autoclaved flask.
  Arms: Intervention Group

SUMMARY:
This research will overview the effect of aloe vera gel (AVG) as intra canal medicament in patients with asymptomatic periapical lesions. It will provide endodontists with scientific evidence regarding the beneficial use of AVG as an intracanal medicament owing to its superior antibacterial and analgesic properties as compared to routinely used commercial intra canal medicaments.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of aloe vera gel based on clinical signs and symptoms as an intracanal medicament in asymptomatic periapical lesions over a period of three weeks. Methodology: Fresh AVG will be prepared. It will be placed as intracanal medicament after cleaning and shaping in patients with asymptomatic periapical lesions in group A while in group B (control group) no intracanal medicament will be placed. Patients will be randomly divided into two groups by randomization in Statistical Package for Social Sciences software (SPSS v24.0). They will be recalled for one week and three week follow ups and in case of no clinical signs and symptoms endodontic procedure will be completed. Statistical analysis: Descriptive statistics will be used for reporting age. Frequencies and percentages will be calculated for categorical variables and intergroup comparison will be done by chi square test

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients presenting with asymptomatic periapical lesions in permanent teeth

Exclusion Criteria:

* History of allergy to AVG

  * Comorbidities likely to impair healing
  * Pregnant women
  * History of previous endodontic treatment in the same tooth
  * Presence of pulp calcification
  * Internal or external root resorption

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Presence or absence of signs and symptoms of the patient | One week and 3 weeks
  Patients in both the groups will be recalled after one week. They will be assessed clinically for either presence or absence of signs and symptoms.
  1. In cases of absence of clinical signs and symptoms, endodontic treatment will be completed.
  2. In cases where patient returns with presence of clinical signs and symptoms, dressing will be removed, and canals will be irrigated with sodium hypochlorite followed by saline. After drying the canals, in group A, AVG will be placed in the canals and tooth restored temporarily while in group B, cotton pellet will be placed in the canals and tooth restored temporarily. The patients will be recalled after two weeks.
  3. If a patient reports with acute symptomsin either of the groups, the protocols to manage acute infection will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Azam, BDS,FCPS, Principal Investigator — Islamabad Dental Hospital
Locations (1):
- Islamabad Dental Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No